CLINICAL TRIAL: NCT04196829
Title: Comparative Evaluation of Staining Potential and Caries Arresting Effect of Silver Diamine Fluoride⁄Potassium Iodide and Silver Diamine Fluoride in Carious Primary Anterior Teeth
Brief Title: Staining Potential and Caries Arresting Effect of Silver Diamine Fluoride⁄Potassium Iodide and Silver Diamine Fluoride
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohsen Aly, lecturer in pediatric dentistry and dental public health, faculty of dentistry, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDF staining potential
Record Dates: First submitted 2019-12-08; First posted 2019-12-12 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silver diamine fluoride ⁄ potassium Iodide (Experimental): 38% silver diamine fluoride and a saturated solution of potassium iodide
  Interventions: Drug: silver diamine fluoride ⁄ potassium Iodide
- silver diamine fluoride (Active Comparator): 38% silver diamine fluoride
  Interventions: Drug: Silver Diamine Fluoride

INTERVENTIONS:
Drug: silver diamine fluoride ⁄ potassium Iodide — The affected tooth surface will be gently cleaned and dried with cotton gauze. The gingival tissue of the tooth will be protected with petroleum jelly. An applicator will be dipped into the SDF and 3-4 mg applied to the lesion with microbrush which will be used to paint solution over carious lesion then we will wait for 1 minute till absorption . Then after SDF application KI will be applied using a separate microbrush which will be saturated by the solution and will be used to paint solution over carious lesion , no rinse will be performed and special instructions will be given following application
  Other Names: SDF / KI
  Arms: silver diamine fluoride ⁄ potassium Iodide
Drug: Silver Diamine Fluoride — The affected tooth surface will be gently cleaned and dried with cotton gauze. The gingival tissue of the tooth will be protected with petroleum jelly. An applicator will be dipped into the SDF and 3-4 mg applied to the lesion with microbrush which will be used to paint solution over carious lesion then we will wait for 1 minute till absorption .
  Other Names: SDF
  Arms: silver diamine fluoride

SUMMARY:
the main objective of this study is to evaluate staining potential and Caries Arresting Effect of silver diamine fluoride⁄potassium Iodide and silver diamine fluoride in carious anterior primary teeth

DETAILED DESCRIPTION:
Despite increased attention on caries prevention, not all children receive preventive treatments and large numbers still experience tooth decay. Primary care providers have had little option other than invasive and costly specialist treatment in the hospital under general anesthesia. In this context, there is interest in simple treatments to halt progress of carious lesions after tooth decay onset. Among these simple treatments is silver diamine fluoride (SDF) treatment. The major drawback to SDF treatment has been its black staining, which has limited its use. To counter the staining, researchers have tested SDF treatment immediately followed with application of saturated solution of potassium iodide (KI).

ELIGIBILITY:
Inclusion Criteria:

* Children with carious primary anterior teeth.
* Children with no spontaneous pain

Exclusion Criteria:

* Tooth mobility
* Signs of pulpal or periapical infection
* Severe medical conditions that would not allow management in the clinic
* Sensitivity to silver or other heavy-metal ions
* Presence of any gingival or perioral ulceration or stomatitis

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
staining potential | base line and Immediately after material application
  change in color of carious lesion using spectrophotometer with unit of measurement percent

SECONDARY OUTCOMES:
caries arresting effect | 3 months, 6 moths, 9 months, 12 months
  evaluating hardness of carious lesion by tactile examination using probe, binary (soft or hard)

OTHER OUTCOMES:
post operative pain | 3 months, 6 moths, 9 months, 12 months
  asking the patient, Binary (present or absent)

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Aly, Phd, Principal Investigator — Lecturer, Faculty of Dentistry, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt